CLINICAL TRIAL: NCT04329468
Title: Detachable String Magnetically Controlled Capsule Endoscopy for Complete Examination of Upper Gastrointestinal Tract and Small Bowel
Brief Title: Detachable String MCE for Upper Gastrointestinal Tract and Small Bowel
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhuan Liao (Other)
Responsible Party: Sponsor-Investigator, Zhuan Liao, Clinical Professor, Changhai Hospital
Organization: Changhai Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: DS-MCE-UGI and SB
Record Dates: First submitted 2020-03-27; First posted 2020-04-01 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-03

CONDITIONS: Capsule Endoscopy
Keywords: DS-MCE; Z-line; Duodenal papilla; Completion rate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DS-MCE examination (Experimental): Subjects with or without digestive symptoms will be enrolled to take DS-MCE and conventional esophagogastroduodenoscopy (EGD) within 48h successively.
  Interventions: Device: DS-MCE

INTERVENTIONS:
Device: DS-MCE — The subjects swallowed the MCE to investigate the esophagus repeatedly by pulling up or down the string. After completion of the esophageal examination, MCE reached the stomach and was lifted away from the posterior wall, rotated if necessary and advanced to the fundus and cardiac regions, and then to the gastric body, angulus, antrum and pylorus. After finishing the stomach examination, the capsule would enter the duodenum due to peristalsis when the pylorus opened. Then DS-MCE tried to inspect the duodenum repeatedly under the string and magnetic field control, including view of major papilla in the descending part of duodenum and retrograde view of pylorus in duodenal bulb with a "360-degree automatic scanning" mode. After completion of the duodenum examination, the capsule started to view the small bowel.

SUMMARY:
This study aims to evaluate the feasibility and safety of DS-MCE with a novel way for complete examination in UGI tract and small bowel, compared with EGD.

DETAILED DESCRIPTION:
Magnetically controlled capsule endoscopy (MCE) has been widely used in clinical practice for upper gastrointestinal (UGI) tract and Small Bowel. However, the complete visualization of UGI tract still present challenges due to rapid transit through esophagus and duodenum, although technical improvements of MCE are helpful.

Detachable String MCE (DS-MCE) can control the movement of MCE through the string and MCE can start next examination after string detachment, which was proved to be an effective and safe method for complete viewing of the esophagus and stomach. In order to improve the duodenum visualization, endoscopist separate MCE from the string after finishing UGI examination so that can inspect the esophagus, stomach and duodenum under the string and magnetic field control.

This is a prospective, single-centered, self-controlled pilot study. Subjects with or without digestive symptoms receiving UGI endoscopy will be enrolled to take DS-MCE and conventional esophagogastroduodenoscopy (EGD) within 48h successively.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients aged 18 to 80
2. With or without gastrointestinal complaints
3. Scheduled to undergo a capsule endoscopy for both stomach and small bowel
4. Signed the informed consents before joining this study

Exclusion Criteria:

1. Pacemakers or electromedical devices implanted which are incompatible with magnetic field;
2. Suspected or known gastrointestinal stenosis, obstruction or other known risk factors for capsule retention;
3. Scheduled magnetic resonance imaging examination before excretion of capsule;
4. Pregnancy or suspected pregnancy;
5. Any contraindications about EGD.
6. Other circumstances that doctors consider inappropriate for the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2020-03-10 (Actual); Primary Completion 2020-08-20 (Estimated); Study Completion 2020-09-20 (Estimated)

PRIMARY OUTCOMES:
Success rate of UGI and small-bowel examination | up to 2 weeks
  The feasibility of DS-MCE examination with a novel way is evaluated by the technical success rate, a composite outcome including the successful separation of the string and MCE, repeat viewing of esophagus, stomach and duodenum, and complete small-bowel examination.

SECONDARY OUTCOMES:
Diagnostic accuracy | up to 2 weeks
  The diagnostic accordance rate, sensitivity and specificity of lesions detected by DS-MCE compared with EGD.
Safety of DS-MCE procedure: presence of any adverse events during DS-MCE procedure will be recorded | up to 2 weeks
  The presence of any adverse events during DS-MCE procedure will be recorded.
Detection rate of Z-line, duodenal papilla and pyloric retrograde view | up to 2 weeks
  The detection means that at least one image of anatomical structure was obtained.
Circumferential visualization of the Z-line and duodenal papilla | up to 2 weeks
  It is defined by quadrants as follows: less than 2 quadrants (< 50%) observed; at least 2 quadrants (50%-75%) observed; at least 3 quadrants (>75%) observed; and entire structure (100%) observed.
Cleansing level of Z-line and duodenal papilla area | up to 2 weeks
  The effect of bubbles/saliva on the appearance of the Z line or duodenal papilla area was both scored as follows: 0=no interference by bubbles/saliva;1=minor interference of bubbles/saliva; 2=major interference of bubbles/saliva.
Visualization level of stomach | up to 2 weeks
  Visualization level of gastric primary anatomic landmarks: cardia, fundus, body, angulus, antrum and pylorus. (good, >75% of mucosa was observed; moderate, 50% to 75% was observed; poor, <50% of the gastric mucosa was observed)
Examination time of esophagus, stomach, duodenum and small bowel | up to 2 weeks
  Record the time taken to finish examination in different digestive part.
Pyloric transit time | up to 2 weeks
  Record the time from completion of the gastric examination to the capsule entering the duodenum.
Discomfort scores associated with DS-MCE | up to 2 weeks
  Discomfort caused by the string, swallowing the DS-MCE, pulling the capsule up or down, and pulling the string out were on a scale from 0 to 3 (0=none;1=mild/minimal; 2=moderate; and 3=severe/very difficult) according to the Ramirez system. Overall discomfort was scored on a scale of 0 to 10 (0=no discomfort; 10=the overall discomfort of EGD) according to our previous system.
Image quality scores | up to 2 weeks
  Assess Image quality grade ranged from 1 to 10 (1, the worst quality; 10, the quality of the best image captured by EGD).
Detection rate of lesions | up to 2 weeks
  The detection rate of lesions in different digestive part (esophagus, stomach, duodenum, jejunoileum) found by MCE.

CONTACTS AND LOCATIONS:
Overall Officials: Zhuan Liao, Study Director — Changhai Hospital, Shanghai, China
Locations (1):
- Changhai Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen YZ, Pan J, Luo YY, Jiang X, Zou WB, Qian YY, Zhou W, Liu X, Li ZS, Liao Z. Detachable string magnetically controlled capsule endoscopy for complete viewing of the esophagus and stomach. Endoscopy. 2019 Apr;51(4):360-364. doi: 10.1055/a-0856-6845. Epub 2019 Mar 1. PMID 30822803
- [Derived] Jiang B, Qian YY, Wang YC, Pan J, Jiang X, Zhu JH, Qiu XO, Zhou W, Li ZS, Liao Z. A novel capsule endoscopy for upper and mid-GI tract: the UMGI capsule. BMC Gastroenterol. 2023 Mar 16;23(1):76. doi: 10.1186/s12876-023-02696-5. PMID 36927462